CLINICAL TRIAL: NCT01999699
Title: A Phase 1 Systems Biology Study to Investigate Immune Correlates of the Response to an Experimental Hepatitis B Vaccine (HEPLISAV) in Healthy Adults 50 to 70 Years of Age.
Brief Title: A Study of the Immune Response to Heplisav in Healthy Older Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dynavax Technologies Corporation (Industry)
Collaborators: Baylor Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: DV2-HBV-22
Record Dates: First submitted 2013-11-26; First posted 2013-12-03 (Estimated); Last update posted 2019-03-20 (Actual); Status verified 2019-03

CONDITIONS: Hepatitis B
Keywords: Heplisav
MeSH Terms: conditions — Hepatitis B | interventions — Hepatitis B Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- HEPLISAV (Experimental)
  Interventions: Biological: HEPLISAV

INTERVENTIONS:
Biological: HEPLISAV

SUMMARY:
This study will investigate the response of the immune system to a hepatitis B (HB) vaccine in healthy adults 50 to 70 years of age. This study is partially funded by the National Institute of Allergy and Infectious Diseases.

DETAILED DESCRIPTION:
The purpose of this study is to examine how the immune system responds to vaccination with HEPLISAV.

ELIGIBILITY:
Inclusion Criteria:

* 50 to 70 years of age, inclusive
* In good health in the opinion of the principal investigator, based upon medical history and physical examination
* Serum negative for HBsAg, anti-HBs, antibody to hepatitis B core antigen (anti-HBc), hepatitis C virus (HCV), and human immunodeficiency virus (HIV)
* If female of childbearing potential, agree to consistently use a highly effective method of birth control from the screening visit through Week 12/Visit 10

Exclusion Criteria:

* Pregnant, breastfeeding, or planning a pregnancy
* Known history of an autoimmune disease
* Previously received any hepatitis B vaccine (approved or investigational)
* Body-mass index (BMI) >30 kg/m2, diabetes mellitus (type 1 or 2), or other chronic medical condition that in the opinion of the principal investigator might interfere with the immune response to hepatitis B vaccination

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2013-11; Primary Completion 2015-02 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Evaluate the changes in cellular responses and gene expression patterns in serial blood samples collected from healthy older adults after vaccination with HEPLISAV. | Day 1, 3, and 7 and on Day 28
Determine which of these changes correlate with the development of protective levels of antibody (anti-HBs >/= 10 milli-international unit (mIU)/mL) to hepatitis B virus (HBV). | Day 1, 3, and 7 and on Day 28

CONTACTS AND LOCATIONS:
Overall Officials: Robert Janssen, MD, Study Director — Dynavax Technologies Corporation
Locations (1):
- Johnson County Clinical Trials, Lenexa, Kansas, United States

IPD SHARING:
Plan to Share IPD: Undecided
a/o August 2016, decision still pending.

REFERENCES:
- See also: Related Info — http://www.dynavax.com